CLINICAL TRIAL: NCT07107555
Title: SnapNSTI: An International Time-bound Prospective Observational Cohort Study Addressing the Epidemiology and Management of Necrotizing Soft Tissue Infections
Brief Title: Necrotizing Soft Tissue Infections
Acronym: SnapNSTI
Status: Enrolling by invitation | Type: Observational
Sponsor: European Society for Trauma and Emergency Surgery (Other)
Collaborators: University of Pennsylvania (Other); Hospital del Mar Research Institute (IMIM) (Other); Hospital del Mar (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); University of Birmingham (Other)
Responsible Party: Principal Investigator, Ana María González Castillo, Principal Investigator, European Society for Trauma and Emergency Surgery
Other Study IDs: SnapNSTI
Record Dates: First submitted 2025-07-25; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Necrotizing Soft Tissue Infection; Fournier Gangrene; Sepsis; Surgical Infection; Soft Tissue Infections
Keywords: diagnosis; management; microbiology; patient related outcome measures; outcomes; NSTI; Necrotizing Soft Tissue Infection; Fournier Gangrene; Soft Tissue Infection; Severe Skin and Soft Tissue Infection; Debridement; Sepsis; Snapshot Audit
MeSH Terms: conditions — Fournier Gangrene; Sepsis; Soft Tissue Infections; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Necrotizing Soft Tissue Infection: This is a prospective, multicenter, observational cohort study of adults (≥18 years) with necrotizing soft-tissue infection (NSTI), defined by surgical/histopathological confirmation or imaging evidence of fascial gas. Participants receive standard care; no interventions are mandated. Data collection includes timing and extent of debridement, antimicrobial regimens, and adjunctive therapies (e.g., intravenous immunoglobulin, hyperbaric oxygen, negative pressure wound therapy), as well as critical care support. Primary outcome is 90-day all-cause mortality; secondary outcomes include organ failure-free days, complications, and 90-day patient-reported outcome measures (PROMs) using EQ-5D-5L. Subgroup analyses will examine variations in practice and outcomes (e.g., immunocompromised status, Fournier's gangrene).

SUMMARY:
SnapNSTI is an international, multicenter, time-bound prospective observational cohort study designed to characterize current epidemiology, management patterns, and outcomes of patients with necrotizing soft-tissue infections (NSTI). The primary objective is to estimate 90-day all-cause mortality and to evaluate the variability in management across centers. The study will also explore the association between clinical characteristics, treatments, and patient-reported outcomes.

DETAILED DESCRIPTION:
Necrotizing soft-tissue infections (NSTIs) are life-threatening surgical emergencies with high mortality despite timely surgical debridement and antibiotic treatment. Wide variability in treatment strategies-ranging from diagnostic imaging to operative timing and adjunctive therapies-contributes to outcome heterogeneity, yet no standardized, high-resolution prospective data exist to guide best practices.

SnapNSTI is a time-bound, multicenter international observational cohort study coordinated by the Center for Emergency Surgery Outcomes Research (CESOR) at the University of Pennsylvania, and led by a consortium of international surgical societies. The study will enroll adult patients with confirmed NSTI over a 6-month window at each participating site within a 12-month period starting in 2026.

The primary outcome is 90-day all-cause mortality. Secondary outcomes include organ support-free days, in-hospital complications, length of stay, and 60-day patient-reported outcomes (PROMs, including the EuroQol 5-Dimension 5-Level (EQ-5D-5L) instrument). Standardized definitions and real-time REDCap-based data collection will ensure data quality. Analyses will include multivariable regression, propensity score methods, and target trial emulation. Results will inform future interventional research and evidence-based guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosis of necrotizing soft-tissue infection (NSTI) confirmed by:

  * Surgical or histopathological evidence of fascial necrosis
  * OR imaging showing gas in the fascial plane
* Admitted to a participating hospital during the enrollment period

Exclusion Criteria:

* Non Severe soft-tissue infection
* Patients <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years or older admitted to participating hospitals with a confirmed diagnosis of necrotizing soft-tissue infection (NSTI). The diagnosis must be based on surgical or histopathological evidence of fascial necrosis, or radiologic confirmation (e.g., gas in the fascial plane). Patients will be enrolled consecutively over a 6-month window at each site. The study includes diverse international centers in all over the world.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
90-day all-cause mortality | 90 days from admission
  All-cause mortality measured at 90 days from hospital admission in patients with confirmed necrotizing soft-tissue infection (NSTI). Mortality status will be obtained via chart review, clinical follow-up or telephone contact.

SECONDARY OUTCOMES:
Organ failure-free days within first 30 days | 30 days from admission
  Number of days alive and free from mechanical ventilation, vasopressors, or renal replacement therapy within 28 days from admission.
Hospital and ICU length of stay | From admision to ICU to discharge to the ward or death
  Number of days from hospital admission to discharge in ICU, including both days. Reported in days, as a continuous variable.
Number and type of reoperations | From admission to 90 days
  Number and type of surgical re-interventions performed after the initial debridement, including amputations, repeat debridement, and drainage procedures.
Patient-reported quality of life (EQ-5D-5L) | 60 days from admission
  Self-reported health status at 60 days after admission using the EuroQol 5-Dimension 5-Level (EQ-5D-5L) instrument. This includes five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain is scored on a 5-point scale (1 = no problems; 5 = extreme problems). The score varies from 5 to 25 points.
Readmission and return to surgery within 90 days | 90 days from admission
  Incidence and reasons for hospital readmissions or return to operating room within 90 days from index admission.

CONTACTS AND LOCATIONS:
Overall Officials: Gary A Bass, MD PhD, Study Chair — University of Pennsylvania; Ana Maria González Castillo, MD PhD, Principal Investigator — Hospital del Mar
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including clinical variables and patient-reported outcomes (PROMs), will be available upon reasonable request and approval by the study Steering Committee.
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 months after publication of primary results, and for a period of 5 years.
Access Criteria: Researchers must submit a methodologically sound proposal to the Steering Committee. Approved proposals will require a data use agreement to ensure appropriate use and protection of data.